CLINICAL TRIAL: NCT03774823
Title: Clinical Evaluation of the Safety and Efficacy of RF and PEMF for the Treatment of Soft Tissue Injury
Brief Title: RF/PEMF Versus Ultrasound for the Treatment of Soft Tissue Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS1217
Record Dates: First submitted 2018-11-26; First posted 2018-12-13 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Soft Tissue Injuries
Keywords: RF/PEMF; Ultrasound
MeSH Terms: conditions — Soft Tissue Injuries | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: One group receives treatment with RF and PEMF while the second group receives treatment with ultrasound
Who Masked: Participant
Masking Description: Participant is not aware which group they will be randomized into upon entering the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Freeze Plus (Experimental): Subjects in this arm will receive treatment using RF and PEMF
  Interventions: Device: RF and PEMF
- Ultrasound (Experimental): Subjects in this arm will receive treatment using ultrasound
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: RF and PEMF — RF and PEMF treatment is deployed using either a small or large handpick applied to the skin and moved slow random patterns homogeneously over the area of treatment
  Arms: Freeze Plus
Device: Ultrasound — Ultrasound is applied to the subject by placing a probe on the treatment area and moving it rapidly and homogeneously over the treatment area
  Arms: Ultrasound

SUMMARY:
The study will investigate whether the impact of PEMF and RF therapies is safe and efficacious for the treatment of pain associated with soft tissue injuries as compared to treatment with ultrasound, and to show the effects of PEMF and RF therapies on range of motion and blood flow associated with soft tissue injuries as compared to ultrasound therapy.

DETAILED DESCRIPTION:
This is a randomized, controlled study of the safety and efficacy of a radiofrequency (RF) and pulsed electromagnetic fields (PEMF) device compared to ultrasound (US) for the treatment of pain associated with soft tissue injuries, and to show the comparative effects on blood flow (BF) and range of motion (ROM). Total expected duration of the clinical study is approximately 6 months (enrollment period of 4 months and a follow-up period of 3 weeks) while individual participation will take three weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and provide written informed consent to receive treatment.
2. Healthy, adult male or female, 18 - 75 years of age.
3. Sustained recent (within 30 days), painful unilateral mild to moderate soft tissue injury.
4. Seeking treatment for pain associated with mild to moderate soft tissue injury.
5. BMI score is greater than 18.5 and less than 29.9.
6. Able and willing to comply with the treatment and follow-up schedule and requirements.

Exclusion Criteria:

1. Pregnant, planning to become pregnant or nursing during the ocurse of the study.
2. Open wound or infection at site of soft tissue injury.
3. Evidence of severe injury, including fracture or nerve injury.
4. History of musculoskeletal disorders, including arthritis, tendonitis, bursitis, ankylosing spondylitis.
5. Moderate to severe ligament tear.
6. Having a known anti-coagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of anticoagulant use as per the subject's physician discretion is permitted).
7. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
8. Having an anesthetic or corticosteroid injection within 4 weeks of study enrollment.
9. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
10. Having a permanent implant in the treated areas, such as metal plates and screws or an injected chemical substance.
11. History of any form of cancer or pre-malignancy in the treatment area.
12. Severe concurrent conditions, such as cardiac disorders, uncontrolled hypertension, etc.
13. Patients with history of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area.
14. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).
15. Poorly controlled endocrine disorders, such as diabetes.
16. Skin piercings in the treatment area.
17. Having a history of anxiety-depression syndromes.
18. Any condition which in the opinion of the investigator may jeopardize the patient's safe participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Biro, Study Director — Venus Concept
Locations (1):
- Kendall Sports Medicine and Rehabilitation Clinic, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Freeze Plus | Ultrasound
Started | 5 | 5
Completed | 4 | 4
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Subjects seeking treatment for pain associated with mild to moderate soft tissue injury.
Groups:
- Total: Total of all reporting groups
Arm/Group | Freeze Plus | Ultrasound | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8
Brief Pain Inventory (Short Form) [Mean (Standard Deviation); unit: score on a scale] — The Brief Pain Inventory - Short Form (BPI-SF) is a self-administered questionnaire made up of the response to 2 components: a) BPI-SF Severity which is the severity of a patient's pain and b) BPI-SF Interference which is the impact of this pain on daily functioning. The patient is asked to rate severity and interference on a 10-point scale where 0 represents 'No pain/No interference' and 10 represents 'Pain/Interference as bad as you can imagine'.
  score on a scale
    BPI-SF Severity | 6.56 (1.72) | 4.38 (2.06) | 5.47 (1.54)
    BPI-SF Interference | 4.75 (2.82) | 0.86 (0.62) | 2.81 (2.75)

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction in BPI-SF Severity
Description: Reduction in pain severity during daily activity at Visit 4 compared to Baseline as measured by the Brief Pain Inventory (Short Form) - Severity. BPI-SF assesses pain at its 'worst', 'least', 'average', and 'now' (current pain) and is rated on a scale of 0-10, where 0 represents 'No pain' and 10 represents 'Pain as bad as you can imagine'.
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 4 | 4
score on a scale | 2.75 (1.86) | 2.44 (1.76)

2. Primary Outcome: Mean Reduction in BPI-SF Interference Score
Description: Reduction in pain interference during daily activity at Visit 4 compared to Baseline as measured by the BPI-SF Interference score. BPI-SF Interference score measures how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. The 0-10 scale is also used for pain interference, where 0 represents 'does not interfere' and 10 represents 'completely interferes'. BPI pain interference is typically scored as the mean of the seven interference items.
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 4 | 4
score on a scale | 2.11 (2.96) | 0.25 (0.96)

3. Primary Outcome: Short Term Blood Perfusion
Description: Change in tissue blood perfusion (BP) pre- and post-treatment at Baseline, Visit 3 as measured by perfusion imaging, measured in perfusion units (PU) where a positive value indicates an increase in blood perfusion and a negative value indicate a decrease in blood perfusion.
Time Frame: Day 8
Population: One subject in the Freeze Plus arm and one subject in the Ultrasound arm did not have blood perfusion measured at visit 3.
Measure: Mean (Standard Deviation); unit: Perfusion units
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 3 | 3
Perfusion units | 21.04 (2.62) | -0.46 (6.38)

4. Primary Outcome: Long Term Blood Perfusion
Description: Change in tissue blood perfusion (BP) pre- and post-treatment at Baseline, Visit 6 as measured by perfusion imaging as measured by perfusion imaging, measured in perfusion units (PU) where a positive value indicates an increase in blood perfusion and a negative value indicate a decrease in blood perfusion.
Time Frame: Day 14
Population: One subject in the Freeze Plus arm and one subject in the Ultrasound arm did not have blood perfusion measured at visit 6.
Measure: Mean (Standard Deviation); unit: Perfusion units
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 3 | 3
Perfusion units | 19.43 (6.13) | 1.44 (4.24)

5. Secondary Outcome: Mean Reduction in BPI-SF Severity Score
Description: Reduction in pain severity during daily activity at Visit 6 as measured by the BPI-SF Severity score. BPI-SF Severity score assesses pain at its 'worst', 'least', 'average', and 'now' (current pain) and is rated on a scale of 0-10, where 0 represents 'No pain' and 10 represents 'Pain as bad as you can imagine'.
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 4 | 4
score on a scale | 2.81 (1.34) | 0.94 (0.94)

6. Secondary Outcome: Mean Reduction in BPI-SF Interference Score
Description: Reduction in pain interference during daily activity at Visit 6 as measured by the BPI-SF Interference score. BPI-SF Interference score measures how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. The 0-10 scale is also used for pain interference, where 0 represents 'does not interfere' and 10 represents 'completely interferes'. BPI pain interference is typically scored as the mean of the seven interference items.
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 4 | 4
score on a scale | 1.43 (1.05) | 0.68 (1.01)

7. Secondary Outcome: Early Subject Satisfaction: 5-Point Likert Satisfaction Scale
Description: Subjects' assessment of satisfaction with the treatment at Visit 4 as measured with a scale, called a 5-point Likert Subject Satisfaction Scale. The scale parameters are defined as:
  4 being very satisfied 3 being satisfied 2 having no opinion
  1 being unsatisfied 0 being very unsatisfied
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 4 | 4
score on a scale | 3.5 (0.6) | 3.5 (1)

8. Secondary Outcome: Midpoint Subject Satisfaction: 5-Point Likert Satisfaction Scale
Description: Subjects' assessment of satisfaction with the treatment at Visit 6 as measured with a scale, called a 5-point Likert Subject Satisfaction Scale. The scale parameters are defined as:
  4 being very satisfied 3 being satisfied 2 having no opinion
  1 being unsatisfied 0 being very unsatisfied
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 4 | 4
score on a scale | 4 (0) | 3.5 (1)

9. Secondary Outcome: Final Subject Satisfaction: 5-Point Likert Satisfaction Scale
Description: Subjects' assessment of satisfaction with the treatment at Visit 7 as measured with a scale, called a 5-point Likert Subject Satisfaction Scale. The scale parameters are defined as:
  4 being very satisfied 3 being satisfied 2 having no opinion
  1 being unsatisfied 0 being very unsatisfied
Time Frame: Day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 4 | 4
score on a scale | 3.4 (0) | 3.5 (1)

10. Secondary Outcome: Assessment of Discomfort
Description: Subject's assessment of discomfort and pain with treatment as measured by a 10 cm visual analog scale (VAS). A line which ranges from 10 being the worst pain ever to 0 being no pain at all.
Time Frame: Day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 4 | 4
score on a scale | 3.025 (.95) | 0.8 (0.27)

11. Secondary Outcome: Adverse Events
Description: Subjects experiencing a treatment-related adverse event (AE)
Time Frame: Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Freeze Plus | Ultrasound
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse data were collected for up to 21 days.
Arm/Group | Freeze Plus | Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT03774823/Prot_SAP_000.pdf